CLINICAL TRIAL: NCT02594748
Title: The Effects of Self-management Education Based on Theory of Planned Behavior on Self-management and Quality of Life of Patients With Type 2 Diabetes and the Other Influencing Factors of Quality of Life
Brief Title: The Effects of Self-management Education Based on Theory of Planned Behavior on Patients With Type 2 Diabetes
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The voluntary attendance rate for intervention is low.
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, FangFang Zhao, PhD student, University of Turku
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BK2014011
Record Dates: First submitted 2015-10-27; First posted 2015-11-03 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental group (Experimental): Intervention is administered to patients in this Arm. The intervention is self-management education based on the theory of planned behavior(TPB). The intervention of experimental group is individual guide and face to face education based on TPB.
  Interventions: Behavioral: Self-management education
- Comparison group (Active Comparator): The comparison group will receive routine care
  Interventions: Behavioral: Routine care

INTERVENTIONS:
Behavioral: Self-management education — The intervention group will receive diabetes self-management education based on the idea of extended theory of planned behavior .
  Arms: Experimental group
Behavioral: Routine care — They will attend the routine lecture in hospital sit and listen, usually 1-2 times during one week in hospital
  Arms: Comparison group

SUMMARY:
The aims of the study are as follows:

* To improve self-management intention and behavior of patients with type 2 diabetes (T2 DM).
* To promote patients to make plans for their self-management and gradually integrate the self-management plan into their daily life.
* To improve resilience, well-being, fatigue and quality of life of patients with T2 DM

In order to achieve the aims, we have set the following objectives:

* To develop and apply self-management education program based on the extended theory of planned behavior.
* To evaluate the efficacy of the educational program:

  1. Self-management education program delivered face to face (intervention group); (b) standard usual care (comparison group).

DETAILED DESCRIPTION:
This study employs a quasi-experimental study design with an intervention and comparison group and follow-up of 3 months; there will be two measuring points (baseline and 3 months after the intervention) , and 9 measures.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥18 years
2. duration of type 2 diabetes ≥3 months
3. without any severe complication and impaired cognition.

Exclusion criteria are:

1. severe physical handicap or mental illness
2. presence of other serious disease such as cancer and stroke.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Audit of Diabetes Dependent Quality of Life at 3-month follow up. | baseline and at three months.
  Measure the impact and important of 19 life domains.

SECONDARY OUTCOMES:
Change from baseline in Fatigue-14 scale at 3-month follow up. | Baseline,3-month follow up.
Change from baseline in Well-Being Index (WHO-5) | Baseline,3-month follow up.
Change from baseline in The Summary of Diabetes Self-Care Activities Measure at 3-month follow up. | Baseline,3-month follow up.
  The scale include diet, exercise, medication, foot care and blood sugar monitoring
Change from baseline in self-management planned behavior developed according to guideline at 3-month follow up. | Baseline,3-month follow up.
  It is based on theory of planned behavior according to the following guideline. Including attitude, subjective norm, perceived behavior control, intention and behavior, action planning and coping planning.The response used likert 1-7 format.
Change from baseline in Connor-Davidson Resilience Scale-10 at 3-month follow up. | Baseline,3-month follow up.
Change from baseline in HbA1c at 3-month follow up. | Baseline, 3-month follow up.
  HbA1c will be measured at outpatient of hospital.
Change from baseline in BMI at 3-month follow up. | Baseline,3-month follow up.
  BMI will be measured at hospital and participants' home.
Change from baseline in Blood sugar at 3-month follow up. | Baseline,3-month follow up.
  Blood sugar will be measured at hospital and participants' home.

CONTACTS AND LOCATIONS:
Overall Officials: Helena leino-kilpi, PhD, Study Chair — Department of Nursing Science, Universtiy of Turku
Locations (1):
- The First People Hospital, Affiliated hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhao FF, Suhonen R, Katajisto J, Stolt M, Leino-Kilpi H. Association between diabetes-related self-care activities and positive health: a cross-sectional study. BMJ Open. 2019 Jul 9;9(7):e023878. doi: 10.1136/bmjopen-2018-023878. PMID 31289048